CLINICAL TRIAL: NCT02619877
Title: Phase 2 Clinical Study to Evaluate Efficacy and Safety of ALLO-ASC-DFU in Patients With Diabetic Foot Ulcers: A Randomized, Comparator-controlled, Single-blind, Parallel-group, Multi-center Study
Brief Title: Clinical Study to Evaluate Efficacy and Safety of ALLO-ASC-DFU in Patients With Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALLO-ASC-DFU-201
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2015-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALLO-ASC-DFU (Experimental): Allogeneic mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-DFU
- Standard therapy (Active Comparator): Standard therapy for patients with diabetic foot ulcer
  Interventions: Other: Standard therapy

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU sheet to diabetic foot ulcer
  Other Names: Allogeneic mesenchymal stem cells
  Arms: ALLO-ASC-DFU
Other: Standard therapy — Standard therapy conducted for patients with diabetic foot ulcer
  Arms: Standard therapy

SUMMARY:
This is a phase II single-blinded study to evaluate the efficacy and safety of ALLO-ASC-DFU in patients with Diabetic Foot Ulcer, compared to standard therapy.

DETAILED DESCRIPTION:
ALLO-ASC-DFU is a hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells. Adipose-derived stem cells have anti-inflammatory effect and release growth factors such as vascular endothelial growth factor (VEGF) and hepatocyte growth factor (HGF), which can enhance wound healing and regeneration of new tissue, finally may provide a new option in treating a Diabetic Foot Ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 years and 80 years of age.
2. Subject is diagnosed with Type I or Type II diabetes, and had defined as diabetic foot ulcers presence of wound for more than 4 weeks at the screening visit.
3. Ulcer located the foot, and ulcer size is between 1 cm^2 and 25 cm^2.
4. Ulcer extends into the dermis, subcutaneous tissue, tendon or joint capsule (Wagner grade 1 or 2).
5. Ulcer is free of necrotic debris.
6. Subjects had adequate circulation to ulcer as documented by one of the methods below:

   * Palpation of pulses around ulcer using Doppler exam
   * Ankle Brachial index (ABI) values ranging between 0.7 and 1.3, or
   * Transcutaneous Oxygen Pressure (TcPO2) > 30 mmHg.
7. Subject is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Ulcer is of non-diabetic pathophysiology.
2. The ulcer has increased or decreased in size by 30% or more during one week after the screening visit.
3. Subject is Human Immunodeficiency Virus (HIV) positive.
4. Subjects with severe hepatic deficiencies.
5. Subjects with a glycated hemoglobin A1c (HbA1c) level of > 15%.
6. Subject who are allergic or have a hypersensitive reaction to bovine-derived proteins or fibrin glue.
7. Subjects requiring intravenous (IV) antibiotics to treat the index wound infection.
8. Subjects with severe renal deficiencies that is uncontrolled by dialysis
9. Subjects who are pregnant or breast-feeding.
10. Subjects who are unwilling to use an "effective" method of contraception during the study.
11. Current evidence of severe infection including pus drainage from the wound site.
12. Subjects who have a clinically relevant history of alcohol or drugs abuse.
13. Subject's blood sugar is > 450 mg/dL at postprandial.
14. Subjects who are not able to understand the objective of this study or to comply with the study requirements.
15. Subjects who are considered to have a significant disease which can impact the study by the investigator.
16. Subjects who are considered not suitable for the study by the investigator.
17. Subjects who have a history of surgery for malignant tumor within the last five years (except carcinoma in situ).
18. Subjects who are currently or were enrolled in another clinical study within 60 days of screening.
19. Subjects who have undergone wound treatments with cell therapy, dermal substitutes, or other biological therapies within the last 30 days.
20. Subjects who are receiving oral or parenteral corticosteroids, immunosuppressive, or cytotoxic agents to unstable dosage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Proportion of re-epithelialization | During 8 weeks

SECONDARY OUTCOMES:
Proportion of re-epithelialization | During 12 weeks
Time to re-epithelialization | During 12 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Follow up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Kyu Han, MD. PhD., Principal Investigator — Korea University Guro Hospital; Ki-Won Young, MD. PhD., Principal Investigator — Eulji General Hospital; Hyun-suk Suh, MD. PhD., Principal Investigator — Asan Medical Center; Jin Woo Lee, MD. PhD., Principal Investigator — Severance Hospital
Locations (4):
- South Korea (4):
  - Korea University Guro Hospital, Guro-gu, Seoul
  - Eulji General Hospital, Nowon-Gu, Seoul
  - Severance Hospital, Seodaemun-Gu, Seoul
  - Asan medical center, Songpa-Gu, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moon KC, Suh HS, Kim KB, Han SK, Young KW, Lee JW, Kim MH. Potential of Allogeneic Adipose-Derived Stem Cell-Hydrogel Complex for Treating Diabetic Foot Ulcers. Diabetes. 2019 Apr;68(4):837-846. doi: 10.2337/db18-0699. Epub 2019 Jan 24. PMID 30679183